CLINICAL TRIAL: NCT01287221
Title: Double-Blind, Placebo-Controlled Study of Rifampicin in Multiple System Atrophy
Brief Title: Study of Rifampicin in Multiple System Atrophy
Acronym: MSA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: DSMB recommended stopping the study after an interim analysis of the primary endpoint revealed that futility criteria were met.
Sponsor: Phillip Low (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Vanderbilt University (Other); Rare Disease Research Network Autonomic Consortium (Unknown)
Responsible Party: Sponsor-Investigator, Phillip Low, MD, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10-003108; P01NS044233 (NIH); U54NS065736 (NIH)
Record Dates: First submitted 2011-01-28; First posted 2011-02-01 (Estimated); Results first posted 2014-03-28 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-02

CONDITIONS: Multiple System Atrophy
MeSH Terms: conditions — Multiple System Atrophy | interventions — Rifampin; isoniazid, pyrazinamide, rifampin drug combination; Riboflavin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rifampicin (Active Comparator): Subjects randomized to this arm will receive 300 mg Rifampicin two times a day for 12 months.
  Interventions: Drug: Rifampicin
- Placebo (Placebo Comparator): Subjects randomized to this arm will receive placebo capsules twice daily for 12 months. The capsules will contain riboflavin (vitamin B2).
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Rifampicin — 300 mg, 2 times daily
  Other Names: Rifampin; Rifadin; Rimactane; Rifater; Rimactazid; Rimycin; Rofact
  Arms: Rifampicin
Drug: placebo — placebo
  Other Names: vitamin B2; riboflavin
  Arms: Placebo

SUMMARY:
The purpose of this study was to determine whether Rifampicin was effective in slowing or reversing the progression of multiple system atrophy (MSA). Research studies indicate that there is an abnormality in protein synthesis and structure in parts of the brain responsible for MSA (protein misfolding) and the drug Rifampicin could potentially prevent or reverse this protein alteration. The study was done on participants with early MSA. The study consisted of taking the drug 2 times a day for 12 months. Participants underwent an evaluation of symptoms and function and will underwent a neurologic examination at the beginning of the study, at 6 months and at 12 months. They were also be contacted at 3 and 9 months by telephone. Studies were done at 10 participating sites.

DETAILED DESCRIPTION:
MSA is a progressive, fatal disorder characterized by autonomic failure and parkinsonism and/or cerebellar involvement. Neuropathologically, MSA is characterized by glial cytoplasmic inclusions (GCI) of abnormally aggregated α-synuclein (α-syn). This was a study to test the hypothesis that Rifampicin, because of its ability to inhibit the formation of α-synuclein fibrils and disaggregate fibrils already formed, will delay progression or reverse neurologic and autonomic functions and symptoms in MSA. This approach has been proposed as a potential approach to treat parkinsonism and specifically, MSA. In an experimental model of MSA, it was hypothesized that Rifampicin would improve behavioral abnormalities of MSA and halt or reverse the pathological changes. The primary objective was to undertake a double-blind placebo-controlled clinical trial on the effect of Rifampicin on progression of neurological and autonomic failure in MSA.

The Data Safety Monitoring Board (DSMB) recommended stopping the study after an interim analysis of the primary endpoint revealed that futility criteria were met.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 30-80 years old with a diagnosis of Possible or Probable MSA of the parkinsonian subtype (MSA-P) or cerebellar subtype (MSA-C) according to The Gilman Criteria (2008).
* Participants who are less than 4 years from the time of documented MSA diagnosis.
* Participants with an anticipated survival of at least 3 years in the opinion of the investigator.
* Participants who are willing and able to give informed consent.
* "Normal" cognition as assessed by Mini-Mental State Examination (MMSE). We will require a value >24.
* Patients should be able to swallow capsules whole.

Exclusion Criteria:

* Pregnant or lactating females.
* Unified Multiple System Atrophy Rating Scale (UMSARS) score >17 on modified UMSARS I (question 11 eliminated).
* Participants with a clinically significant or unstable medical or surgical condition that, in the opinion of the investigator, might preclude safe completion of the study or might affect the results of the study. These include conditions causing significant Central Nervous System (CNS) or autonomic dysfunction, including congestive heart failure, recent (<6 months) myocardial infarct, thrombocytopenia (<50 x10(9)/L), immunosuppressed state, severe uncontrolled hypertension, severe cardiopulmonary disease, severe anemia (<8g/dl), severe liver or kidney disease (creatinine >2.3 mg/dl) uncontrolled diabetes mellitus (HbA1c >10g%), alcoholism, malignant neoplasms, amyloidosis, uncontrolled hypothyroidism, unstable peripheral neuropathies, concurrent infections, orthopedic problems that compromise mobility and activity of daily living, severe cerebrovascular accidents (such as hemiplegia, aphasia and non-dominant parietal lobe syndrome), and neurotoxins or neuroactive drug exposure, parkinsonism due to drugs (including neuroleptics, a-methyldopa, reserpine, metoclopramide).
* Participants who have taken any investigational products within 60 days prior to baseline.
* Women of child-bearing potential who do not practice an acceptable method of birth control. Acceptable methods of birth control in this study are: surgical sterilization, intrauterine devices, partner's vasectomy, a double-protection method (condom or diaphragm with spermicide), hormonal contraceptive drug (i.e., oral contraceptive, contraceptive patch, long-acting injectable contraceptive) with a required second mode of contraception.
* Participants taking Tetrabenazine, Rasagiline or Selegiline. The participant will qualify for the Rifampicin study after they have stopped these drugs for 3 months
* Participants known to have porphyria.
* Participants with abnormal liver function tests defined as 1.5 times the upper limit of normal.
* Concomitant therapy with anticholinergic, alpha and beta adrenergic antagonists, or other medications that affect autonomic function will be stopped prior to autonomic evaluation.
* The regular use of neuroleptics within the six months prior to the initial evaluation. Occasional use of a neuroleptic as an anti-emetic in the past is allowed, providing not more than three doses were taken within the previous 12 months.
* Since Rifampicin has significant drug-drug interactions, particular attention has been devoted to the use of concomitant medications. Considering the target population, we will exclude participants taking antifungal medication (itraconazole), antiarrhythmics like amiodarone, digitalis and lorcainide, female hormones and quetiapine (Seroquel). Use of methylphenidate, cinnarizine, reserpine, amphetamine, atypical antipsychotics such as risperidone, olanzapine, and quetiapine or a Monoamine oxidase A (MAO-A) inhibitor within one month prior to the baseline visit are also exclusionary.
* Diseases with features of Parkinson's Disease; e.g., progressive supranuclear palsy, essential tremor, inherited cerebellar degeneration, or postencephalitic parkinsonism.
* Dementia (DSM-IV criteria - Amer. Psych. Association, 1994). The score on the MMSE must be >24.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-03; Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip A Low, MD, Principal Investigator — Mayo Clinic; David Robertson, MD, Principal Investigator — Vanderbilt University; Sid Gilman, retired, MD, Principal Investigator — University of Michigan
Locations (10):
- United States (10):
  - UCLA Medical Center, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - Mayo Clinic, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - Harvard Medical School, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - New York University, New York, New York
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Result] Low PA, Robertson D, Gilman S, Kaufmann H, Singer W, Biaggioni I, Freeman R, Perlman S, Hauser RA, Cheshire W, Lessig S, Vernino S, Mandrekar J, Dupont WD, Chelimsky T, Galpern WR. Efficacy and safety of rifampicin for multiple system atrophy: a randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2014 Mar;13(3):268-75. doi: 10.1016/S1474-4422(13)70301-6. Epub 2014 Feb 5. PMID 24507091

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 10 specialized tertiary centers in the United States from April 2011 through April 2012.
Period: Overall Study
Arm/Group | Rifampicin | Placebo
Started | 50 | 50
Completed 3 Months Follow-up | 49 | 50
Completed 6 Months Follow-up | 47 | 43
Completed 9 Months Follow-up | 42 | 40
Completed 12 Months Follow-up | 40 | 39
Completed | 46 | 45
Not Completed | 4 | 5
Not completed — Lack of Perceived Benefit | 1 | 1
Not completed — Adverse Event | 3 | 3
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rifampicin | Placebo | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (7.8) | 61.1 (9.2) | 61.0 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 16 | 39
  Male | 27 | 34 | 61
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100
Multiple System Atrophy (MSA) Type [Number; unit: participants]
  Parkinsonian (MSA-P) | 19 | 22 | 41
  Cerebellar (MSA-C) | 31 | 28 | 59
Certainty of Multiple System Atrophy (MSA) Diagnosis [Number; unit: participants] — Criteria for probable MSA:1)Autonomic failure involving urinary incontinence or an orthostatic decrease of blood pressure within 3 min of standing by at least 30 mm Hg systolic or 15 mm Hg diastolic and 2)Poorly levodopa-responsive parkinsonism, or 3) cerebellar syndrome (gait ataxia with cerebellar dysarthria, limb ataxia, or cerebellar oculomotor dysfunction).
  Criteria for possible MSA:1)Parkinsonism or 2)cerebellar syndrome and 3)at least one feature suggesting autonomic dysfunction (unexplained urinary urgency, frequent bladder emptying, erectile dysfunction, orthostatic hypotension.)
  participants
    Probable | 31 | 34 | 65
    Possible | 19 | 16 | 35

OUTCOME MEASURES:

1. Primary Outcome: Rate of Change From Baseline to 12 Months in the Total Unified Multiple System Atrophy Rating Scale (UMSARS) Part I Score (Minus Question 11)
Description: UMSARS is a scale measuring disease progression that comprises 4 parts; only Parts I and II were used in this study. Part I scores symptoms of neurological and autonomic dysfunction. Part II is a motor examination. Part I has 12 questions with a rating scale ranging from 0 (normal) to 4 (extreme dysfunction). Therefore the total score for Part I could range from 0 (normal) to 48 (extreme dysfunction).
  Participant-specific rate of change in points per month was estimated using slope estimate from least square regression where for each participant, their UMSARS I scores were plotted over time measured in months.
Time Frame: baseline, 12 months
Population: Analysis was done using intention to treat principles and no imputations were done for any missing values or slope estimates. All randomized participants who took at least two doses of the study drug were included in the principal efficacy analysis. One subject on the Rifampicin arm did not return after the baseline visit.
Measure: Mean (Standard Deviation); unit: units on a scale per month
Arm/Group | Rifampicin | Placebo
Number analyzed (Participants) | 49 | 50
units on a scale per month | 0.5 (0.7) | 0.5 (0.5)
Statistical Analysis 1: Comparison: Rifampicin vs Placebo; Given that there were no imbalances identified between the two groups at baseline and the slope estimates for the two treatment arms did not support assumption of normality, the analysis was performed using Wilcoxon rank-sum test; Test type: Superiority or Other; p = 0.82, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change From Baseline to 12 Months in UMSARS Part I Score (Minus Question 11)
Description: UMSARS is a scale measuring disease progression that comprises 4 parts, only Parts I and II were used in this study. Part I scores symptoms of neurological and autonomic dysfunction. Part II is a motor examination. Part I has 12 questions with a rating scale ranging from 0 (normal) to 4 (extreme dysfunction). Therefore the total score for Part I could range from 0 (normal) to 48 (extreme dysfunction).
Time Frame: baseline, 12 months
Population: Analysis was done using intention to treat principles. Not all patients reached the 12 month time point due to missed visits or the early termination of the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rifampicin | Placebo
Number analyzed (Participants) | 39 | 39
units on a scale | 6.2 (5.6) | 5.6 (5.0)
Statistical Analysis 1: Comparison: Rifampicin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.62, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change From Baseline to 12 Months in UMSARS Part II
Description: UMSARS is a scale measuring disease progression that comprises 4 parts; only Parts I and II were used in this study. Part I scores symptoms of neurological and autonomic dysfunction. Part II is a motor examination. Part II has 14 items with a rating scale ranging from 0 (normal) to 4 (extreme dysfunction). Therefore the total score for Part II could range from 0 (normal) to 56 (extreme dysfunction).
Time Frame: baseline, 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rifampicin | Placebo
Number analyzed (Participants) | 36 | 36
units on a scale | 7.0 (6.3) | 5.4 (6.6)
Statistical Analysis 1: Comparison: Rifampicin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.23, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change From Baseline to 12 Months in Total UMSARS (i.e., UMSARS Part I Minus Question 11 + UMSARS Part II)
Description: UMSARS is a scale measuring disease progression that comprises 4 parts; only Parts I and II were used in this study. Part I scores symptoms of neurological and autonomic dysfunction. Part II is a motor examination. Part I has 12 questions with a rating scale ranging from 0 (normal) to 4 (extreme dysfunction). Part II has 14 items with a rating scale ranging from 0 (normal) to 4 (extreme dysfunction). Therefore the total score for total UMSARS Parts I minus Question 11 + Part II could range from 0 (normal) to 104 (extreme dysfunction).
Time Frame: baseline, 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rifampicin | Placebo
Number analyzed (Participants) | 36 | 36
units on a scale | 12.9 (10.6) | 10.8 (10.7)
Statistical Analysis 1: Comparison: Rifampicin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.31, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Rate of Change From Baseline to 12 Months in Total UMSARS (i.e., UMSARS Part I Minus Question 11 + UMSARS Part II) Using Slope Estimate
Description: UMSARS is a scale measuring disease progression that comprises 4 parts; only Parts I and II were used in this study. Part I scores symptoms of neurological and autonomic dysfunction. Part II is a motor examination. Part I has 12 questions with a rating scale ranging from 0 (normal) to 4 (extreme dysfunction). Part II has 14 items with a rating scale ranging from 0 (normal) to 4 (extreme dysfunction). Therefore the total score for total UMSARS Parts I minus Question 11 + Part II could range from 0 (normal) to 104 (extreme dysfunction).
  Participant-specific rate of change in points per month was estimated using slope estimate from least square regression where for each participant, their total UMSARS scores were plotted over time measured in months.
Time Frame: baseline, 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale per month
Arm/Group | Rifampicin | Placebo
Number analyzed (Participants) | 45 | 43
units on a scale per month | 1.1 (1.0) | 1.2 (1.2)
Statistical Analysis 1: Comparison: Rifampicin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.65, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change From Baseline to 12 Months in the COMPASS-Select Scale
Description: The composite autonomic symptoms score (COMPASS) provides a score of autonomic symptom severity with appropriate weighting. In the COMPASS_select, symptoms are confined to 6 select domains of symptoms. The version of the COMPASS-Select used (06-09-2009 v1) has 46 questions, with multiple parts, scores ranging from "much worse" to "no such symptoms." Scores could range from 0 (no such symptoms) to 85 (much worse).
Time Frame: baseline, 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rifampicin | Placebo
Number analyzed (Participants) | 39 | 38
units on a scale | 6.9 (16.5) | 4.6 (13.4)
Statistical Analysis 1: Comparison: Rifampicin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.61, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Change in the COMPASS-Select-Change Scale From Baseline to 12 Months
Description: The change in COMPASS is a derivative of COMPASS and evaluates the change in symptoms over time on selected domains of symptoms as a function of natural history or intervention therapy. The focus is on 7 selected domains. The version of the COMPASS-Change -Select Scale used (06-09-2009 Ver. 1) has 16 questions, with multiple parts, scores ranging from "much worse" to "no such symptoms." The score could range from 0 (no such symptoms) to 94 (much worse).
Time Frame: baseline, 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rifampicin | Placebo
Number analyzed (Participants) | 39 | 38
units on a scale | 41.4 (33.8) | 32.1 (35.7)
Statistical Analysis 1: Comparison: Rifampicin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.22, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were to be recorded from the time a participant signed the informed consent form and throughout the 12 months of the study, even if they prematurely discontinued the study drug.
Description: The attribution of serious adverse events was determined by the Medical Review Officer, whereas the attribution of non-serious adverse events was determined by the reporter.
Arm/Group | Rifampicin | Placebo
Serious Adverse Events (participants affected / at risk) | 3/50 | 12/50
Other Adverse Events (participants affected / at risk) | 31/50 | 26/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rifampicin (N=50) | Placebo (N=50)
Joint Function (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Infection with unknown ANC (Infections and infestations) | 1 (1) | 0 (0)
Musculoskeletal/soft tissue - other (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Thrombosis/thrombus/embolism (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac ischemia/infarction (Cardiac disorders) | 0 (0) | 1 (1)
Vessel injury - artery (Cardiac disorders) | 1 (1) | 0 (0)
Death not associated with CTCAE Term (Cardiac disorders) | 0 (0) | 2 (2) — 2 subjects died post-study, unrelated to study drug or placebo.
Mood Alteration (Psychiatric disorders) | 0 (0) | 1 (1)
Cardiac general - other (Cardiac disorders) | 0 (0) | 1 (1)
Renal/genitourinary - other (Renal and urinary disorders) | 0 (0) | 1 (2)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Liver Dysfunction/failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Obstruction/stenosis of airway (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neurology - other (Nervous system disorders) | 0 (0) | 1 (1)
Vomiting - aspirated/stroke (Vascular disorders) | 0 (0) | 1 (1) — Subject hospitalized for hernia repair surgery, and surgery went well. Subject was being cleaned by family and vomited, aspirated, and stroked. Subject experienced multiple system failure and was declared dead.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rifampicin (N=50) | Placebo (N=50)
Speech impairment (General disorders) | 0 (0) | 1 (1)
Prolonged QTc Interval (Cardiac disorders) | 0 (0) | 1 (1)
Leukocytes (Immune system disorders) | 1 (1) | 0 (0) — Total White Blood Count (WBC)
Nausea (Gastrointestinal disorders) | 6 (6) | 1 (1)
Neutrophils/granulocytes (Immune system disorders) | 1 (1) | 0 (0) — Absolute neutrophil count (ANC)/Absolute granulocyte count (AGC)
Wound complication, non-infectious (Infections and infestations) | 0 (0) | 1 (1)
Renal/Genitourinary - Other (Renal and urinary disorders) | 3 (4) | 8 (12)
Urinary frequency/urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 6 (6) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 3 (3) | 2 (2)
Petechiae/purpura (Vascular disorders) | 1 (1) | 0 (0) — hemorrhage/bleeding into skin or mucosa
Edema: limb (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Infection with unknown (Infections and infestations) | 2 (2) | 1 (4) — ANC
Lymphopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Eyelid dysfunction (Eye disorders) | 0 (0) | 1 (1)
Glucose, serum-low (Endocrine disorders) | 0 (0) | 1 (1) — hypoglycemia
Constitutional Symptoms - other (General disorders) | 0 (0) | 3 (3)
Creatinine (Renal and urinary disorders) | 1 (1) | 3 (3)
Neurology - other (Nervous system disorders) | 4 (4) | 5 (5)
Ataxia (Nervous system disorders) | 0 (0) | 2 (2) — lack of voluntary coordination of muscle movements
Nasal Cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Cystitis (Renal and urinary disorders) | 2 (2) | 0 (0)
Gastrointestinal - other (Gastrointestinal disorders) | 5 (5) | 4 (4)
Musculoskeletal/soft tissue - other (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Taste Alteration (dysgeusia) (General disorders) | 1 (1) | 0 (0)
Tremor (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 1 (1) | 0 (0)
Vision - photophobia (Eye disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 3 (4) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 1 (1) — (including neurogenic bladder)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (General disorders) | 0 (0) | 2 (2)
Urine color change (Renal and urinary disorders) | 5 (5) | 6 (6)
Hemorrhage/bleeding - other (Vascular disorders) | 1 (1) | 2 (2)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Metabolic/Laboratory - other (General disorders) | 4 (5) | 4 (8)
Syncope (fainting) (General disorders) | 1 (1) | 1 (1)
Endocrine - other (Endocrine disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Allergic reaction/hypersensitivity (General disorders) | 0 (0) | 1 (1) — (including drug fever)
Blood/Bone marrow - other (Vascular disorders) | 1 (1) | 1 (1)
Dysphagia (difficulty swallowing) (General disorders) | 0 (0) | 1 (1)
Glucose, serum-high (Endocrine disorders) | 0 (0) | 2 (2) — (hyperglycemia)
Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hepatobiliary/Pancreas - other (Endocrine disorders) | 1 (1) | 1 (1)
Joint Function (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rigors/chills (General disorders) | 0 (0) | 1 (1)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary/Upper Respiratory - other (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2)
Sweating (diasporesis) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Mood alteration (Psychiatric disorders) | 1 (1) | 0 (0)
Weight loss (General disorders) | 1 (1) | 0 (0)
Vision - blurred vision (Eye disorders) | 1 (1) | 0 (0)
Bone: spine - scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Somnolence/depressed level of consciousness (General disorders) | 0 (0) | 1 (1)
Dermatology/Skin - other (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 1 (1) | 0 (0)
Obstruction/stenosis of airway (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
International Normalized Ratio (INR) of prothrombin time (Vascular disorders) | 0 (0) | 1 (1)
ALT, serum glutamic pyruvic transaminase (SGPT) (Hepatobiliary disorders) | 1 (1) | 2 (6)
AST, serum glutamic oxaloacetic transaminase (SGOT) (Hepatobiliary disorders) | 0 (0) | 1 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dry mouth/salivary gland (xerostomia) (General disorders) | 1 (1) | 0 (0)
Memory Impairment (Psychiatric disorders) | 0 (0) | 1 (1)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 2 (2) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
CNS cerebrovascular ischemia (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated early; the Data Safety and Monitoring Board recommended stopping the study after an interim analysis of the primary endpoint revealed that futility criteria were met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No